CLINICAL TRIAL: NCT03173209
Title: Evaluating the Effectiveness of the Calm Moments Cards Program Implemented by School Personnel
Acronym: CMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FY2016-49
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Stress; Child, Only
Keywords: school

STUDY DESIGN:
Intervention Model Description: A one-group (N 93) mixed-methods design using a pretest-posttest survey and qualitative analysis of written reﬂections was used to explore the meaning and outcomes of the Calm Moments Cards program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- school professional development (Other): Professional development in Calm Moments Cards program. Occupational therapists used lecture and coaching to educate school personnel on signs of stress and how to embed evidence based strategies (cognitive behavioral, mindfulness, and sensory) throughout the school day to reduce stress and enhance emotional well-being in students using the Calm Moments Cards program.
  Interventions: Behavioral: professional development in Calm Moments Cards program

INTERVENTIONS:
Behavioral: professional development in Calm Moments Cards program — Professional development (lecture and coaching)was used in combination with informal coaching by occupational therapy practitioners to educate school personnel on signs of stress and how to embed evidence based strategies (cognitive behavioral, mindfulness, and sensory) throughout the school day to reduce stress and enhance emotional well-being in students using the Calm Moments Cards program.

SUMMARY:
We explored the meaning and outcomes of a 4-month program designed to build capacity of school personnel in implementing evidence-based strategies for reducing stress and promoting mental well-being among students in school settings. A one-group (N 93) mixed-methods design using a pretest-posttest survey and qualitative analysis of their written reactions was used to explore the meaning and outcomes of the Calm Moments Cards program.

DETAILED DESCRIPTION:
In order to explore the effectiveness of the Calm Moments Cards program on school personnel's ability to recognize signs of stress and the implementation of embedded strategies to reduce stress and enhance emotional well-being, we conduct a mixed-methods research study using pretest-posttest surveys (assessing knowledge, beliefs, and actions) and qualitative analysis of written reflections about the meaning and use of the Calm Moments Cards. The focus of the intervention is on prevention of stress and anxiety based on situational stressors (e.g. taking a test, completing an assignment) so that students can focus on and succeed in doing their schoolwork. Occupational therapy practitioners oriented school personnel to the signs of stress and the use of the 17 Calm Moments Cards using a 1 hour inservice. This was followed by informal coaching to foster implementation.

ELIGIBILITY:
Inclusion Criteria:

* School personnel representing teachers, related service providers and para-educators working with elementary students in schools

Exclusion Criteria:

* School personnel who were informed of but declined to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-01-17 (Actual); Primary Completion 2016-10-13 (Actual); Study Completion 2016-10-13 (Actual)

PRIMARY OUTCOMES:
Change in knowledge, beliefs, and actions regarding recognizing and reducing stress in children | 4 months
  20 questions using Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Susan Bazyk, PhD, Principal Investigator — Cleveland State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Calm Moments Cards — http://www.everymomentcounts.org
- Available data/document: intervention materials: Calm Moments Cards program — http://www.everymomentcounts.org — Calm Moments Cards program